CLINICAL TRIAL: NCT02656368
Title: Safety and Efficacy of SEBORRHEAMEDIS Face Cream in Patients With Seborrheic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamedis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAM-SEB_FC-01
Record Dates: First submitted 2016-01-06; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-03

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional, open label, Safety/Efficacy Study (Experimental): SEBORRHEAMEDIS Face Cream Interventional 30
  Interventions: Device: SEBORRHEAMEDIS Face Cream

INTERVENTIONS:
Device: SEBORRHEAMEDIS Face Cream — SEBORRHEAMEDIS Face Cream is a barrier-based, non-steroidal cream. The cream includes plant extracts The cream was designed to manage the symptoms of facial Seborrheic dermatitis symptoms such as erythema, scaling and pruritus.

SUMMARY:
SEBORRHEAMEDIS Face Cream is a barrier-based, non-steroidal cream. The cream includes plant extracts The cream was designed to manage the symptoms of facial Seborrheic dermatitis symptoms such as erythema, scaling and pruritus.

DETAILED DESCRIPTION:
30 subjects will be enrolled to the study. After eligibility is confirmed, subjects will be asked to sign an Informed Consent form.

At the baseline visit, the investigator will select a target area on the face. The target area will be evaluated for erythema (redness) and desquamation (scaling) using a 5-point scale: 0 = none, 1 = minimal, 2 = mild, 3 = moderate and 4 = severe. Photography of the target area will be taken. For reference, a fixed object (such as a ruler) will be photographed in the same frame. In addition, the investigator will assess the overall facial lesions using an ISGA based on a 5-point scale. The subject will evaluate his/her pruritis over the past 24 hours, using a 5-point scale: 0 = no itching, 1 = minimal and rare itching, 2= mild itching, (subject is aware of the itching only when relaxed), 3= moderate itching (subject is often aware of the itching, which occasionally disturbs sleep), 4 = severe and constant itching.

Subjects will be instructed to use SEBORRHEAMEDIS Face Cream twice a day, morning and evening, for a consecutive period of 42 days. In addition to the baseline visit (day 0), subjects will be asked to come to the clinic for two follow-up visits at days 14 and 28 and for a final visit at day 42. A flexibility of ±2 days will be allowed. In case of an adverse event, the subject will be asked to immediately contact the clinic, and to come to an unscheduled visit if needed.

At each of the two follow-up visits and at the final visit, the investigator will evaluate the overall severity of seborrhea (ISGA) and the target area's erythema and desquamation. The subject will assess his/her pruritus over the past 24 hours.

At the final visit, the subject will also complete a product-assessment questionnaire. The questionnaire will ask several questions about satisfaction attributes, using a 5-point scale: -2 = very unsatisfied, -1 = unsatisfied, 0 = neutral, +1 = satisfied, +2 = very satisfied. Attributes will include: overall satisfaction, speed of results, ease of use, ease of spread, comfort under makeup, feel on the skin (-2 = very greasy, +2 = very moisturizing), speed of absorption, texture, color and odor

ELIGIBILITY:
Inclusion Criteria:

* Subject with mild (ISGA=2) to moderate (ISGA=3) facial Seborrheic dermatitis.
* Male or female aged 18 years or older.
* Subject who agrees not to use any Seborrheic Dermatitis medication during the study, except for the tested product.
* Subject is willing to sign an Informed Consent

Exclusion Criteria:

* Subject pregnant or lactating.
* Subject has a condition that requires continuous systemic or topical corticosteroid or antimycotic therapy
* Subject has a severe disease that is likely to interfere with the study conducting
* Subject has a known sensitivity to any of the ingredients contained in the tested product.
* Subject is expected to be extensively exposed to the sun during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement of overall ISGA. Descriptive Name of scale. Physician dermatology evaluation. | Days 42

SECONDARY OUTCOMES:
Improvement of erythema, desquamation on the target area. Physiological parameter. Physician dermatology evaluation. | Days 0, 14, 28 and 42
Improvement of pruritus. Physiological parameter. Assessed by subject. | Days 0, 14, 28 and 42
Number and severity of Adverse Events | Days 0, 14, 28 and 42

CONTACTS AND LOCATIONS:
Overall Officials: Rubén del Rio Gil, MD, Principal Investigator — Hospital de l'Esperit Sant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barak-Shinar D, Del Rio R, Green LJ. Treatment of Seborrheic Dermatitis Using a Novel Herbal-based Cream. J Clin Aesthet Dermatol. 2017 Apr;10(4):17-23. PMID 28458770